CLINICAL TRIAL: NCT02022839
Title: B-lines at Lung Ultrasound Predicts Weaning Failure From Mechanical Ventilation
Brief Title: Role of Lung Ultrasound in Predicting Weaning Outcomes
Status: Completed | Type: Observational
Sponsor: Hospital Moinhos de Vento (Other)
Responsible Party: Principal Investigator, Augusto Savi, PhD, Hospital Moinhos de Vento
Other Study IDs: 2010/125
Record Dates: First submitted 2011-04-27; First posted 2013-12-30 (Estimated); Last update posted 2013-12-30 (Estimated); Status verified 2013-12

CONDITIONS: Ventilator Weaning; Ultrasonography
Keywords: mechanical ventilation, weaning; ultrasonography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Days
Oversight: Data Monitoring Committee: No

SUMMARY:
We aimed to verify the potencial role of bedside lung ultrasound findings of critically ill patients candidates to liberation from mechanical ventilation in predicting weaning outcomes. The analysis will be taken in two times: immediately before and at the and spontaneous breathing trial.

ELIGIBILITY:
Inclusion Criteria:

* Invasive mechanical ventilation > 24 hours
* Eligibility to weaning from mechanical ventilation

Exclusion Criteria:

* Tracheostomy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Mechanical ventilation patients in a mixed intensive care unit
Sampling Method: Non-Probability Sample
Enrollment: 250 (Actual)
Dates: Start 2010-12; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Weaning Failure | Participants will be followed up til weaning success or weaning failure at the end of spontaneous breathing trial. In case of weaning success, then they will be followed for more 48 hours to detect extubation failure.

CONTACTS AND LOCATIONS:
Overall Officials: Ana Carolina P Antonio, MD, Principal Investigator — Hospital Moinhos de Vento, Universidade Federal do Rio Grande do Sul; Cassiano Teixeira, MD, PhD, Study Chair — Hospital Moinhos de Vento; Marli Knorst, MD, PhD, Study Chair — Federal University of Rio Grande do Sul
Locations (1):
- Hospital Moinhos de Vento, Porto Alegre, Rio Grande do Sul, Brazil

REFERENCES:
- [Derived] Antonio ACP, Teixeira C, Castro PS, Zanardo AP, Gazzana MB, Knorst M. Usefulness of radiological signs of pulmonary congestion in predicting failed spontaneous breathing trials. J Bras Pneumol. 2017 Jul-Aug;43(4):253-258. doi: 10.1590/S1806-37562016000000360. PMID 29364998
- [Derived] Antonio AC, Teixeira C, Castro PS, Savi A, Oliveira RP, Gazzana MB, Knorst M. 48-Hour Fluid Balance Does Not Predict a Successful Spontaneous Breathing Trial. Respir Care. 2015 Aug;60(8):1091-6. doi: 10.4187/respcare.03172. Epub 2015 Apr 28. PMID 25922544